CLINICAL TRIAL: NCT02786472
Title: ConnectEd: A Randomized Controlled Trial Connecting Through Educational Training
Acronym: ConnectEd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heather Bush (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Heather Bush, Associate Professor, Biostatistics, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC R01CE 2690.1
Record Dates: First submitted 2016-05-20; First posted 2016-06-01 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Sexual Violence
Keywords: Bystander behaviors; Incoming students; CampusSave; Prevention; Sexual Assault; Incapacitation
MeSH Terms: interventions — Convolutional Neural Networks

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Haven (Active Comparator): Online Bystander Training or Haven provides students with definitions and statistics associated with sexual assault and relationship violence, bystander skills and strategies, and campus policies and resources. The trainings are "personalized and reflective" and incorporate the student's "unique perspectives and experiences." This 45-minute training is mandatory and students are asked to complete a follow-up survey 45-days after the training. Because this training is mandatory for all incoming students, all students are expected to have exposure to this training.
  Interventions: Behavioral: Online Bystander Training
- AlcoholEdu (Active Comparator): Online Substance Abuse Training or AlcoholEdu provides confidential substance abuse education course which uses a science-based approach to educate students about alcohol and its effects. Whether the student drinks or not, the course will help them make informed decisions about alcohol and better deal with drinking behavior that may occur around them. AlcoholEdu is used by more than 500 colleges nationwide through EVERFi.
  Interventions: Behavioral: Online Substance Abuse Training
- ConnectEd (Experimental): In-person Combination Training provides Green Dot Intensive Bystander Training AND Substance Abuse Prevention cross-programming to develop ConnectED. The intentional coordination between substance abuse and violence prevention programming would include in-depth information related to interpersonal violence and substance use/abuse, activities to help participants explore their connection to these issues; information and activities related to the culture of violence, drinking and drug use and how everyone has a role in impacting that culture; information about bystander behaviors and barriers to taking action when they encounter problem situations; participant self-evaluation of their own attitudes, beliefs and biases around these issues; and, in-depth skill building activities to prepare participants to safely intervene in problem situations.
  Interventions: Behavioral: In-Person Combination Training
- GreenDot (Experimental): In-person Bystander Training provides Green Dot bystander intervention program (www.livethegreendot.com) seeks to empower potential bystanders (students) to actively engage their peers in violence prevention. Intensive bystander training involves interactive, skill development with role-play of bystander behaviors. This program focuses on building knowledge and skills related to interpersonal violence and being an active bystander. There is a structured curriculum for both introductory sessions and longer, skill-building sessions. While a Popular Opinion Leader strategy has been used in prior training, for this trial all incoming students randomized to this condition will be offered intensive bystander training.
  NOTE: Green Dot Speeches will be supplemental to Intensive Green Dot Bystander training. These speeches will continue to occur as usual. As the aim of this study is to compare bystander intensive training, we will not attempt to limit participation to Green Dot Speeches.
  Interventions: Behavioral: In-Person Bystander Training

INTERVENTIONS:
Behavioral: Online Bystander Training — Large groups of 120-150 students will complete Haven training via computer; training lasts duration of the online program.
  Other Names: Haven
  Arms: Haven
Behavioral: Online Substance Abuse Training — Large groups of 120-150 students will complete EverFi training via computer; training lasts duration of the online program.
  Other Names: AlcoholEdu
  Arms: AlcoholEdu
Behavioral: In-Person Bystander Training — In-person training of large groups of 120-150 students; training lasts 3-4 hours
  Other Names: Green Dot
  Arms: GreenDot
Behavioral: In-Person Combination Training — In-person training of large groups of 120-150 students; training lasts 3-4 hours
  Other Names: ConnectEd
  Arms: ConnectEd

SUMMARY:
The purpose of this randomized intervention pilot is to evaluate the relative efficacy of bystander training elements (delivery mode and integration of substance abuse prevention) among cohorts of incoming undergraduates at the University of Kentucky, a nationally recognized leader in addressing sexual violence through bystander intervention programming. Consenting students will be randomized to one of the following training conditions:

1. In-person Green Dot Intensive Bystander-based Sexual Violence Prevention Training (GreenDot);
2. In-person Green Dot Intensive Bystander Training combined with Substance Abuse Prevention Training;
3. Online Bystander-based Sexual Violence Prevention Training (Haven), and;
4. Online Substance Abuse Training (AlcoholEdu).

DETAILED DESCRIPTION:
Rates of sexual violence (SV) or dating violence (DV) remain high among college students (22% in the past year for female undergraduates). Binge drinking commonly occurs (25% of undergraduates report binge drinking in the past month) and is a strong predictor of sexual risk taking and violence victimization and perpetration. Given connections between SV/DV risk and alcohol use and abuse, many advocate prevention programming to jointly address SV/DV and alcohol abuse. Bystander interventions, recognized as promising violence prevention strategies, are unique in their engagement of all community members to 1) recognize situations that may become violent and 2) learn to safely and effectively intervene to reduce violence risk. Based on their promise, the Campus Sexual Violence Elimination Act (SaVE) now requires all publicly-funded colleges to provide bystander intervention in the hopes of reducing sexual violence. No randomized intervention trial has compared bystander interventions focused exclusively on SV/DV prevention with those additionally addressing alcohol abuse prevention within the bystander context. We propose such an experimental trial at the University of Kentucky (UK), a nationally recognized leader in addressing sexual violence through bystander intervention programming. The purpose of this randomized intervention trial is to evaluate the relative efficacy of bystander training elements. In this study will be randomized to one of the following: 1) Online Bystander Training (Haven), 2) Online Substance Abuse Training (AlcoholEdu), 3) In-person Bystander Training (Green Dot Intensive Training), or 4) In-person Bystander/Substance Abuse Training (ConnectEd). Aim 1: Evaluate methods to capture behaviors and diffusion of training through social media communications (e.g., Facebook, Twitter, Instagram). Aim 2: Determine the relative efficacy of the three bystander training conditions to a) increase bystander efficacy and behaviors by domain (alcohol abuse and violence prevention), b) reduce acceptance of SV/DV, alcohol's role in sexuality, and alcohol use / abuse, and c) reduce risk taking behaviors by domains of sexual behavior and alcohol use or abuse. Aim 3: Determine the relative cost of implementing bystander approaches and their cost effectiveness. Design: Incoming UK undergraduates will be recruited and randomized to one of the four conditions and followed for 9 months, one academic year (n=4000, total over 2 academic year cohorts). A mixed-method approach will be used to measure intervention fidelity and costs over time and by condition. Using the most rigorous design available, we seek to generate new understanding of how novel bystander intervention approaches work to reduce not only SV/DV risk taking behaviors but also reduce alcohol abuse.

Incoming students will be invited to participate in a randomized trial testing bystander program efficacy. Those consenting to study participation will be randomized to one of the four conditions. These conditions include:

1. In-person Green Dot Intensive Bystander-based Sexual Violence Prevention Training (GreenDot);
2. In-person Green Dot Intensive Bystander Training combined with Substance Abuse Prevention Training (WellAware);
3. Online Bystander-based Sexual Violence Prevention Training (Haven), and;
4. Online Substance Abuse Training (AlcoholEdu).

All incoming students (17-24) agreeing to study participation will be invited to complete surveys at baseline (prior to training), and at end of the fall and spring semesters. Additionally, students will be asked to complete micro-surveys using the myUK app.

Student recruitment will be conducted as students are entering UK during their summer orientation (June and July). We anticipate that at 45-50% of students will agree to study participation and provide data; thus our final participant pool is expected to consist of 4,000 participants from academic years 2016 and 2017.

Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation, median, first and third quartiles, and min and max); categorical variables will be described with counts and percentages. Change scores and percent change scores will be calculated from baseline (prior to start of first academic year) as well as from end of Fall to Spring within each academic year. Numerical and graphical summaries will be provided overall, by subpopulation within college communities (e.g., by gender, sexual attraction, fraternity/sorority or athletic team membership) and most importantly by training condition. Simple comparisons of groups will be made using ANOVA for continuous variables and chi-square tests for categorical outcomes. Comparisons between groups will be conducted as randomized; simple comparisons of continuous variables between groups will be performed using ANOVA and chi-square tests of independence for categorical variables. Although groups will be randomly assigned, potential confounders will be examined with bivariate analyses and comparisons requiring covariate adjustment will use regression modeling (e.g. ANCOVA, logistic regression). Planned subgroup analyses include analyses by gender group, by sexual attraction, by Greek life participation. These will also be conducted as randomized and as received. Effect modification will also be assessed by including interactions in regression models (linear, logistic, and mixed models depending on outcomes and the presence of longitudinal measures). SAS v9.4 will be used for all data management and statistical analysis; a significance level of 0.01 will be used for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

-Incoming University of Kentucky undergraduate students (2016, 2017)

Exclusion Criteria:

* Any current/non-incoming University of Kentucky student
* Any student primarily enrolled at another college or university

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3178 (Actual)
Dates: Start 2016-05; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of Bystander Behaviors | baseline, 5 months and 9 months
  The primary outcome for this study is bystander behaviors as measured by the number of behaviors reported by students overall and by domain. Bystander behaviors are measured through reports of actual behaviors. These primary bystander behavior outcomes will be used to evaluate the relative efficacy of the intervention(s). As bystander behaviors require opportunity, these primary outcomes will be examined accounting for the presence of opportunity to bystand. The primary analysis will be the comparison of these outcomes over time using mixed models, with a particular interest on whether there is a condition by time interaction (time: baseline, 5 months post, 9 months post).
Change in Bystander Behavior Intentions Scale | baseline, about 5 months and 9 months
  Students will report their intention to engage in bystander behaviors. The scale used to report this is a five point Likert scale. Questions include measures such as, likelihood of becoming involved based on their relation to the individual and likelihood to report based on disciplinary actions. The changes that are measured throughout the academic year will be used to report intentions in bystander behavior.
Change in Bystander Behavior Efficacy Scale | baseline, 5 months and 9 months
  Students will report their self efficacy in their ability to preform bystander behaviors. The scale used to report this efficacy is a five point Likert scale. Questions include measures such as, self reported ability to recognize risky situations and reported skill set of prevention of violence behaviors. The changes that are measured throughout the academic year will be used to report efficacy in bystander behavior.
Count of Bystander Behaviors Engagement with Peers | about 2 months, about 4 months, 5 months, about 7 months, and 9 months
  Students will report bystander behaviors that they participated in with their peers. These are reported using multiple choice and open ended questions to describe the event and the action taken by an individual who engaged in a bystander behavior. Questions include what bystander action was preformed, where the incident occurred, and number of times this event occurred. The number of times students indicate these behaviors will be combined across surveys.

SECONDARY OUTCOMES:
Change in Acceptance of SV/DV Scale | baseline, 5 months and 9 months
  Students will be asked questions that describe their acceptance of sexual violence and dating violence. The scale used to report this acceptance are a five point Likert scale. Questions include measures such as, fights add excitement to a romantic relationship and people who wear revealing clothing are asking for trouble. The changes that are measured throughout the academic year will be used to report change in acceptance of sexual violence and dating violence behaviors.
Count of self-reported risky behaviors, sexual and alcohol related | baseline, 5 months and 9 months
  Students will be asked about frequency of binge drinking, incapacitation, and opportunities to observe high risk situations. The number of times students indicate these behaviors will be combined across follow-up surveys.

OTHER OUTCOMES:
Social media and campus communications (e.g., Twitter, Instagram, Facebook, myUK) | One Academic Year (9 months)
  This is an exploratory outcome to determine potential diffusion of interventions. Students electing to participate in this part of the trial, will have posts and comments aggregated over the study period. Sentiment analysis and word clouds will be used to determine if language from trainings diffuse into social media communications.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Bush, PhD, Principal Investigator — University of Kentucky; Ann L Coker, MPH, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-03-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT02786472/ICF_000.pdf